CLINICAL TRIAL: NCT03709732
Title: Register Research Combined With Health Surveys and Patient Data, to Assess Work Participation and Quality of Life Among Persons With Spinal Cord Injury and Their Caregivers
Brief Title: Living With Spinal Cord Injury.
Status: Completed | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/294
Record Dates: First submitted 2018-10-15; First posted 2018-10-17 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Spinal Cord Injuries
Keywords: Quality of Life; Registries; Norway; Caregivers; Employment
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Spinal cord injury: Persons with a spinal cord injury. No intervention
  Interventions: Other: no intervention
- Caregivers spinal cord injury: Caregivers for persons with a spinal cord injury. No intervention
  Interventions: Other: no intervention
- Controls for patients: Control group for patient cohort. No intervention
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — observational study

SUMMARY:
A Spinal Cord Injury (SCI) often drastically disrupts the lives of affected patients and their relatives and caregivers. This observational study will provide new knowledge on how patients and their family caregivers cope in the first years after injury in terms of work inclusion, participation, care giver burden and quality of life. This project will utilize Norwegian spinal cord injury quality register data and link clinical individual data from the quality register to national administrative data on employment and social insurance benefits.

DETAILED DESCRIPTION:
All individuals in the Norwegian Spinal Cord Injury Registry (NorSCIR) in the period 2011-2017, meaning that they have already given their consent, will be asked to participate. They will be sent a letter with information about the study including a questionnaire.

In the letter they will also be asked, if they agree, to forward an invitation letter to their closest caregiver addressed to "the main family caregiver".

Main family caregiver will be defined as persons who are providing unpaid assistance and support to the person with a SCI. The letter for the caregiver with information about the study, includes a questionnaire. All patients in the NorSCIR and their main caregivers (after consent) will be linked to national administrative register to provide data on social insurance benefits, education and work.

Control groups from the general population will be selected and identified in the national registries (for both the patient cohort and caregiver cohort). These control groups will be used to compare the level of work/benefit over time for patients and caregivers with that of the general population. Also, within-person approaches will be used to assess the impact of the injury, comparing each participant's status in the period after injury with their own status at a time period before injury.

20.04.2022 A relatively low proportion of family caregivers responded to the questionnaire (N = 73). Only 61 gave their consent to link their data to data from Statistics Norway and the Norwegian Labour and Welfare Administration. We had, therefore, to reconsider this part of the project. We have now concluded that the caregiver population is too small to link their information to the national administrative registers and to make a comparison with a control group from the general population. A control group for caregivers was therefore not needed anymore.

ELIGIBILITY:
Cohort 1:

Inclusion criteria:

* registered in the Norwegian spinal cord injury quality registry
* giving informed consent, i.e. accept that the information in the registry (included linked information in national registers)

Exclusion criteria:

* younger than 16 years

Cohort 2:

Inclusion criteria:

* providing unpaid assistance and support to the person with a spinal cord injury
* chosen by the patient.

Exclusion criteria:

* younger than 16 years

Cohort 3 :

Inclusion:

* Control groups from the general population, for patients
* identified in the national registries

Exclusion criteria:

* younger than 16 years

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cohort 1:
  All individuals in NorSCIR in the period 2011-2017, meaning that they have already given their consent, will be asked to participate.
  Cohort 2:
  Main family caregiver will be defined as persons who are providing unpaid assistance and support to the person with a spinal cord injury.
  Cohort 3 :
  A control group from the general population will be selected and identified in the national registries ( the patient cohort).
Sampling Method: Non-Probability Sample
Enrollment: 2654 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Work participation of persons with a spinal cord injury | 2 years
  Before and after injury
Work participation of family caregivers | 2 years
  Before and after their role as a caregiver
Mental Health of patients by MHI-5 | 2 years
  The mental Health is measured with the Mental Health Index (MHI-5)
Quality of life of patients by WHOQoL-5 | 2 years
  QoL is measured with the 5-item World Health Organization Quality of Life Assessment (WHOQoL-5)
Quality of life of patients by ISCI QoL Data set | 2 years
  QoL is measured with the International SCI quality of life Basic Data Set (ISCI QoL Data Set)
Mental health of family caregivers by MHI-5 | 2 years
  Mental health is measured with the Mental Health Index (MHI-5).
Quality of life of family caregivers by WHOQoL-5 | 2 years
  QoL is measured with the 5-item World Health Organization Quality of Life Assessment (WHOQoL-5)
Quality of life of family caregivers by ISCI QoL Data Set | 2 years
  QoL is measured with the International SCI quality of life Basic Data Set (ISCI QoL Data Set)
Caregiver burden by Caregiver strain index | 2 years
  Caregiver burden for family caregivers is measured with the Caregiver strain index
Caregiver burden by Self rated burden scale | 2 years
  Caregiver burden for family caregivers is measured with the Self rated burden scale.
Participation by PAM-13 for patients | 2 years
  Participation is measured with the following instruments: Patient Activation Measure (PAM-13).
Participation by PAM-13 for family caregivers | 2 years
  Participation is measured with the following instruments: Patient Activation Measure (PAM-13)
Participation by Utrecht scale for Evaluation of rehabilitation participation | 2 years
  Participation for patients is measured with the Utrecht Scale for Evaluation of Rehabilitation Participation (USER-P).
Participation by Utrecht scale for Evaluation of rehabilitation participation (adjusted) | 2 years
  Participation for family caregivers is measured with the adjusted Utrecht Scale for Evaluation of Rehabilitation Participation (USER-P).

CONTACTS AND LOCATIONS:
Overall Officials: Johan Skomsvoll, md phd, Study Director — St. Olavs Hospital; Annette Halvorsen, md, Principal Investigator — St. Olavs Hospital
Locations (1):
- St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided